CLINICAL TRIAL: NCT06879028
Title: The Outcome of Various Methods of Surgical Reconstruction of Depressed Skull Fractures
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Islam Mostafa, Islam Mostafa AbdelBary Ebrahim, Assiut University
Other Study IDs: CDAUHNS
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Head Trauma Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cases presented with Depressed Fractures needing surgical intervention at Assiut University Hosppita

SUMMARY:
* To investigate the outcomes of different approaches to surgical repair/Elevation of Traumatic Depressed Skull Fractures
* To improve the outcome of surgical elevation of depressed fractures regarding the rate of post-operative deficit and complications, as well as the aesthetics and patient recovery

DETAILED DESCRIPTION:
Depressed Fractures are of the commonest conditions seen in Head injuries; its incidence is unknown, but it is seen most commonly in Assault by hard objects and Road Traffic Accidents (8) and other high momentum collisions with the skull. Parietal bone is the most commonly fractured, followed by Temporal, Occipital and Frontal bones (1,8) They are classified mainly as Simple (Closed) or Compound (Open). Depressed fractures can be managed conservatively (2,3) but surgical intervention is needed if the depression is greater than calvarium thickness (1,2,8) or the fracture is over the Superior Sagittal Sinus, or risk infection from external debris. (4,6) Depressed Fractures when associated with underlying intracranial pathology (Mostly Haematoma or contusions) (1,2,8) require surgical elevation and management of other complications.

Elevation and debridement is recommended as the surgical method of choice. All management strategies for compound depressed fractures should include antibiotics. (1,2,8) Paediatric populations have better outcome (3,7) due to possibility for future remodelling and cranial growth.

Safe and effective surgical techniques to elevate Depressed fractures include craniotomy, surgical elevation with primary replacement of bone fragments in place, elevation through a burr hole at the periphery, fixation of bone fragments with miniplates, or fixation of bone fragments with vicryl sutures.

However, no available studies signify a preferable approach to depressed fractures or outcome of different methods. So, our study will try to identify and establish a significant treatment plan and preferable approach.

1. Golfinos JG, Cooper PR. Skull fracture and post-traumatic cerebrospinal fluid fistula. In: Head Injury, 4th, Cooper PR, Golfinos JG (Eds), McGraw-Hill, New York 2000. p.155.
2. Bullock, M. R., Chesnut, R., Ghajar, J., Gordon, D., Hartl, R., Newell, D. W., … Wilberger, J. (2006). Surgical Management of Depressed Cranial Fractures. Neurosurgery, 58(Supplement), S2-56-S2-60. doi:10.1227/01.neu.0000210367.14
3. Bonfield, C. M., Naran, S., Adetayo, O. A., Pollack, I. F., & Losee, J. E. (2014). Pediatric skull fractures: the need for surgical intervention, characteristics, complications, and outcomes. Journal of Neurosurgery: Pediatrics, 14(2), 205-211. doi:10.3171/2014.5.peds13414
4. HESHAM EL-SOBKEY, M.D., Ph.D., A. F. K. M. P. Surgical Elevation for Symptomatic Depressed Skull Fractures Over Dural Venous Sinus. The Medical Journal of Cairo University, 2019; 87(June): 1917-1925. doi: 10.21608/mjcu.2019.54048
5. Nnadi MO, Bankole OB, Arigbabu SO. Outcome of surgically treated non-missile traumatic depressed skull fracture. Niger Postgrad Med J. 2014 Dec;21(4):311-4. PMID: 25633449.
6. Abdelaal, M., Saro, A., Fadl, K., Abdelrahman, A. Management of Compound Depressed Fractures Over Major Cranial Venous Sinuses. The Egyptian Journal of Hospital Medicine, 2021; 83(1): 1177-1182. doi: 10.21608/ejhm.2021.161776
7. Al-Haddad SA, Kirollos R. A 5-year study of the outcome of surgically treated depressed skull fractures. Ann R Coll Surg Engl. 2002 May;84(3):196-200. PMID: 12092875; PMCID: PMC2503833.
8. Prakash A, Harsh V, Gupta U, Kumar J, Kumar A. Depressed Fractures of Skull: An Institutional Series of 453 Patients and Brief Review of Literature. Asian J Neurosurg. 2018 Apr-Jun;13(2):222-226. doi: 10.4103/ajns.AJNS_168_16. PMID: 29682012; PMCID: PMC5898083.

ELIGIBILITY:
1. Inclusion criteria:

   1. Any patient of both sexes admitted to Trauma unit with total coverage of 1 year.
   2. Patients with Surgically indicated Depressed Skull Fractures
2. Exclusion criteria:

   1. Patients with congenital causes of depressed fractures 2. Patients with Old trauma (1 month or more). 3. Patients with Severe Polytrauma, and no evident Neurosurgical emergency. 3. Patients that need ICU/ CCU admission. 4. Patients with Expressed Fractures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient of both sexes admitted to Trauma unit.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Rates of Surgical Sites infection | 6 months
Cosmosis and Post Op Appearance | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code